CLINICAL TRIAL: NCT03879304
Title: Effectiveness of a Multimodal Physiotherapy Program With Virtual Reality Glasses in Duchenne and Becker.
Acronym: RVDuchenne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Rosa Baeza Barragán, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UMalagaRV
Record Dates: First submitted 2019-03-09; First posted 2019-03-18 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Muscular Dystrophy, Duchenne and Becker Types
Keywords: Virtual Reality [L01.224.160.875], [L01.296.555]; Physical Therapy Modalities [E02.779], [E02.831.535]; Respiratory Therapy [E02.880]; Dystrophin [D12.776.210.500.250]; Becker Muscular Dystrophy [C10.668.491.175.500.300]; Resistance training [E02.831.535.483.875]; Muscular Stretching Therapy [E02.831.535.483.750]
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Twelve participants were randomized to follow a multimodal physiotherapy program for 6 weeks. At the end of this period the participants will be crossed to another intervention without virtual reality glasses. The results will be measured before and after each intervention during the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal physiotherapy program with RV (Experimental): The RV intervention group receives a tele multimodal physiotherapy program with tradicional exercises of physiotherapy like stretching, aerobic, training through videos and gamification with VR glasses.
  Interventions: Other: multimodal physiotherapy program with RV
- Traditional physiotherapy program (Active Comparator): Traditional intervention group receives assistance of a program of physiotherapy traditional without virtual reality glasses.
  Interventions: Other: traditional physiotherapy program

INTERVENTIONS:
Other: multimodal physiotherapy program with RV — Physiotherapy Programm includes: respiratory physiotherapy, stretching, resistance training, aerobic training and adaptation and training with virtual reality glasses and relaxation.
  Arms: Multimodal physiotherapy program with RV
Other: traditional physiotherapy program — Multimodal physiotherapy Programm includes: traditional physiotherapy, stretching, massage.
  Arms: Traditional physiotherapy program

SUMMARY:
Duchenne's Muscular Dystrophy and Becker Dystrophy, hereafter DMD and BMD, is a serious and progressive disease that affects 1 in 3,500-6,000 males born alive. Scale 6-minute walking test, is used for determine the inclusion of children with DMD in pharmacological studies. Furthemore, is used to verify a training effectiveness assessing muscular endurance and cardio-respiratory functions. This Research evaluates the feasibility and effectiveness of a multimodal physiotherapist program with virtual reality glasses.

DETAILED DESCRIPTION:
In addition a physiotherapy program, virtual reality have a lot of importance advantages for train while motivated the kids.

A cross over study will be applied. In the control time, patient will received a initial evaluation and a final without making the physiotherapy program and without virtual reality glasses. The data will be collected by principal examiner.

In the intervention time the group will received 10 multimodal physiotherapy sessions, two or one per week, along six weeks. Also they are going to training walking with with virtual games.

Multimodal physiotherapist program describes the exercises to be performed, how long it will take, the number of repetitions and the way to do it with the physiotherapist in zoom session.

At the end of the multimodal physiotherapy program, variables will be evaluated by the principal examiner.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 and 15 years
* Duchenne and Becker Diagnosis ICD-10 issued by specialist in neurology.
* Children who can walk 10 m at last 120 seconds.
* First punctuation of North Start Ambulatory assessment bigger than 20 points.

Exclusion Criteria:

* An other Dystrophies.
* Older than 10 years.
* Not Physiotherapy. Not walk.
* Asociated heart disease Sprains, fractures. FC >120, Sat O2 <89%.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in six meter walking test (6-MWT) score | Baseline, up to six weeks
  Six-meter walking test is a a well-established outcome measure in a variety of diseases. It is accurate, reproducible, simple to administer, and well tolerated. The 6MWT is a robust assessment tool for use in clinical trials given its ability to quantitatively evaluate ambulation in a controlled environment.

SECONDARY OUTCOMES:
EPInfant | through study completion, average 6 weeks
  Scale of perceived child effort measurement EPInfant. It shows 11 numerical descriptors (0 to 10), 5 verbal descriptors located every 2 levels of intensity, and a set of illustrations that represent a child running at increasing intensities along a scale of bars of incremental height following a exponential type slope from left to right. The higher value represent a worse outcome.
NSAA o North Star Ambulatory Assessment | Baseline, up to 6 weeks
  Functional scale for children with DMD. It is expressed in points and evidences the acquisition of functions or the loss of them. Whilst DMD children may generally present with recognizable adaptations to activity due to the underlying progressive muscular weakness, they may modify their activity to achieve functional goals in slightly differing ways. Generally, activities are graded in the following manner:
  2 - 'Normal' - no obvious modification of activity
  1 - Modified method but achieves goal independent of physical assistance from another 0 - Unable to achieve independently. The better punctuation is 34 point, what mean the higher outcome.
MFM o Motor Function Measure | Baseline, up to 6 weeks
  measure motor performance
Kids Screen-52 | Baseline.
  quality of life test

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín Valero, PhD, Study Director — Universidad de Málaga; Maria Teresa Labajos Manzanares, PhD, Study Director — Universidad de Málaga
Locations (1):
- Universidad de Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
an average of 2 years

REFERENCES:
- [Background] Baeza-Barragan MR, Labajos Manzanares MT, Ruiz Vergara C, Casuso-Holgado MJ, Martin-Valero R. The Use of Virtual Reality Technologies in the Treatment of Duchenne Muscular Dystrophy: Systematic Review. JMIR Mhealth Uhealth. 2020 Dec 8;8(12):e21576. doi: 10.2196/21576. PMID 33289679
- [Result] Baeza-Barragan MR, Labajos Manzanares MT, Amaya-Alvarez MC, Morales Vega F, Rodriguez Ruiz J, Martin-Valero R. Effectiveness of a 5-Week Virtual Reality Telerehabilitation Program for Children With Duchenne and Becker Muscular Dystrophy: Prospective Quasi-Experimental Study. JMIR Serious Games. 2023 Nov 15;11:e48022. doi: 10.2196/48022. PMID 37990809